CLINICAL TRIAL: NCT01334866
Title: Graft Patency Outcomes in Patients Undergoing Coronary Artery Bypass Grafting Via Minimally Invasive Coronary Surgery
Acronym: MICS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D03782
Record Dates: First submitted 2011-04-05; First posted 2011-04-13 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Arteriosclerosis of Coronary Artery Bypass Graft
Keywords: Minimally invasive coronary surgery; Coronary artery bypass grafting; MICS CABG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Minimally invasive coronary artery bypass graft surgery — The MICS CABG procedure can bridge the gap between percutaneous coronary intervention (PCI) and standard sternotomy. The key components are direct vision, creating anastomoses with traditional instruments and proximal aortic location.
  Other Names: MICS CABG

SUMMARY:
This clinical study has been developed to evaluate the clinical outcomes in patients undergoing coronary artery bypass grafting via Minimally Invasive Coronary Surgery (MICS); a minimally invasive coronary bypass procedure that is done on a beating heart via a smaller chest incision, thus avoiding the invasiveness of the standard procedure.

ELIGIBILITY:
Inclusion Criteria:

* > or equal to 18 and < or equal to 80 years of age
* Suitable minimally invasive coronary surgery (MICS) candidate for non-emergent first time, single or multivessel coronary artery bypass grafting (on pump or off pump)
* Left ventricle ejection fraction >30%
* Willing and able to provide written informed consent and comply with study requirements

Exclusion Criteria:

* Severe cerebrovascular disease within 90 days of surgery including history of prior stroke.
* Previous cardiac surgery procedures such as CABG revisions, surgical ablations or valve replacements
* Congestive heart failure with a New York Heart Association (NYHA) Class IV
* History of renal insufficiency (i.e. prior serum creatinine of >2mg/dl) and/or requiring dialysis
* Uncontrolled diabetes (i.e. >2 serum glucose concentrations of >350 mg/dl)
* Severe uncontrolled systemic hypertension (i.e. systolic pressure >160 mmHg)
* Peripheral/systemic active infection excluding the patient from cardiac surgery
* Life expectancy of less than 1 year due to other illness such as cancer or pulmonary, hepatic or renal disease
* Participation in another investigational protocol that may confound the results of this study
* Female of child bearing potential and lactating or intends to become pregnant during the study
* Severe distal disease and small posterior lateral targets

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McGinn, MD, Principal Investigator — Staten Island University Hospital
Locations (2):
- Staten Island University Hospital, Staten Island, New York, United States
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Ruel M, Shariff MA, Lapierre H, Goyal N, Dennie C, Sadel SM, Sohmer B, McGinn JT Jr. Results of the Minimally Invasive Coronary Artery Bypass Grafting Angiographic Patency Study. J Thorac Cardiovasc Surg. 2014 Jan;147(1):203-8. doi: 10.1016/j.jtcvs.2013.09.016. Epub 2013 Oct 30. PMID 24183338
- See also: Medtronic, Inc. Corporate Website — http://www.medtronic.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 91 subjects were enrolled, with 89 subjects receiving the study treatment. The first subject was enrolled on December 30, 2009 and the last subject was enrolled on October 4, 2012. Of the 89 subjects treated with the study procedure, 72 subjects completed the 6 month follow-up primary endpoint visit.
Groups:
- Minimally Invasive Coronary Artery Bypass Grafting: 91 subjects were enrolled, with 89 subjects receving the study treatment. Of the 89 subjects treated with the study procedure, 72 subjects completed the 6 month follow-up primary endpoint visit.
Period: Overall Study
Arm/Group | Minimally Invasive Coronary Artery Bypass Grafting
Started | 91 (91 subjects were enrolled in the study; with 89 subjects receiving the study treatment.)
Completed | 72
Not Completed | 19
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 3
Not completed — medically necessary prior to procedure | 2
Not completed — medically necessary post-procedure | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Completion Cohort: 91 subjects were enrolled, with 89 subjects receving the study treatment. Of the 89 subjects treated with the study procedure, 72 subjects completed the 6 month follow-up primary endpoint visit.
Arm/Group | Study Completion Cohort
Number analyzed (Participants) | 91
Age Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 81
Region of Enrollment [Number; unit: participants]
  United States | 45
  Canada | 46

OUTCOME MEASURES:

1. Primary Outcome: Technical Success (Graft Patency) in a MICS Approach
Description: For each subject, the endpoint for technical success (graft patency) in a MICS approach is defined as acceptable flow for graft size for an anastamosis. This will be characterized by the surgeon's assessment/angiography after the graft is complete.
Time Frame: At time of procedure (day 1)
Measure: Number; unit: percentage of grafts
Units Other Than Participants: Grafts
Groups:
- Minimally Invasive Coronary Artery Bypass Grafting: 89 Subjects received study treatment
Arm/Group | Minimally Invasive Coronary Artery Bypass Grafting
Number analyzed (Participants) | 89
Number analyzed (Grafts) | 208
percentage of grafts | 100

2. Primary Outcome: Procedural Success in a MICS Approach
Description: A successful procedure can be defined as a procedures not requiring conversion (sternotomy). This will be characterized by whether the graft procedure can be completed through the minimally invasive thoracotomy without having to convert to a sternotomy in order to complete the grafting.
Time Frame: At time of procedure (day 1)
Measure: Number; unit: percentage of subjects
Groups:
- Study Procedure Cohort: 89 Subjects received study treatment
Arm/Group | Study Procedure Cohort
Number analyzed (Participants) | 89
percentage of subjects | 100

3. Primary Outcome: Patency of the Index Graft at 6 Months
Description: For each subject, the endpoint is the percent of stenosis collected on the subject's 6 month angiography form. This will be characterized for each graft using the FitzGibbon scoring system based on the 64-Slice CT Angiography results.
  The FitzGibbon Scoring system is as follows:
  A:Excellent graft with unimpaired runoff (< 50% stenosis) B:Stenosis reducing caliber of proximal or distal anastomoses or trunk to <50% of the grafted coronary artery.
  O:Occluded (100% stenosed)
Time Frame: 6 months post-procedure
Measure: Number; unit: percentage of grafts
Units Other Than Participants: Grafts
Arm/Group | Minimally Invasive Coronary Artery Bypass Grafting
Number analyzed (Participants) | 89
Number analyzed (Grafts) | 165
percentage of grafts
  Grade A | 90.9
  Grade B | 0.6
  Grade O | 8.5

4. Primary Outcome: Composite Major Adverse Event Rate (Early)
Description: During procedure and within 30 days post-procedure or hospital discharge, whichever is longer. The adverse events will include:
  * Major hemorrhage/bleeding requiring surgical intervention
  * Aortic complications
  * Graft vessel revision (GVR)
  * Transient ischemic attacks (TIA)
  * Cerebrovascular accidents (CVA)/stroke
  * Myocardial infarction (MI)
  * Death
Time Frame: During procedure (day 1) and within 30 days post-procedure or hospital discharge, whichever is longer (throughout 6 month evaluation)
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Minimally Invasive Coronary Artery Bypass Grafting
Number analyzed (Participants) | 89
percentage of subjects | 2.2 [0 to 6.9]

5. Secondary Outcome: Composite Major Adverse Event Rate (Late)
Description: Characterize the composite major adverse event rate after 30 days post-procedure or hospital discharge, whichever is longer through the 6-Month evaluation. The major adverse events will include:
  * Major hemorrhage/bleeding requiring surgical intervention
  * Aortic complications
  * Graft vessel revision (GVR)
  * Transient ischemic attacks (TIA)
  * Cerebrovascular accidents (CVA)/stroke
  * Myocardial infarction (MI)
  * Death
Time Frame: After 30 days post-procedure or hospital discharge, whichever is longer through the 6-Month evaluation
Measure: Number; unit: percentage of subjects
Arm/Group | Minimally Invasive Coronary Artery Bypass Grafting
Number analyzed (Participants) | 89
percentage of subjects | 0

ADVERSE EVENTS:
Time Frame: Adverse events reported from treatment through 6-month follow-up.
Description: Adverse events were classified as serious by the PI following ISO 14155 standards.
Arm/Group | Study Procedure Cohort
Serious Adverse Events (participants affected / at risk) | 14/89
Other Adverse Events (participants affected / at risk) | 46/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Procedure Cohort (N=89)
Angina (Cardiac disorders) | 1 (1)
Anemia and blood loss (Blood and lymphatic system disorders) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 3 (3) — Bleeding (2), Bleeding/Oozing (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Low Cardiac Index (Cardiac disorders) | 3 (3) — Low cardiac index (2), low cardiac index and central venous pressure (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical Blood Loss (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Procedure Cohort (N=89)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Atrial Fibrillation (Cardiac disorders) | 15 (15)
Hypertension (Vascular disorders) | 9 (9)
Hypotension (Vascular disorders) | 13 (13)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Subcutaneous Emphysema (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Atelectasis and Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less